CLINICAL TRIAL: NCT06792266
Title: Identification of Possible Circular RNA-MicroRNA-Messenger RNA Regulatory Axis As a Predictor for IVF Outcome
Brief Title: CircularRNA-microRNA-mRNA Regulatory Axis in IVF
Acronym: IVF
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Lamia Ahmed, assisstant lecturer, Assiut University
Other Study IDs: CircularRNA-microRNA-mRNA axis
Record Dates: First submitted 2025-01-15; First posted 2025-01-24 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-01

CONDITIONS: Infertility (IVF Patients)
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — follicular fluid samples from a single follicle >18 mm will be collected and centrifuged at 1500×g for 15 min to separate the serum fraction debris; the supernatant will be stored at -80 °C for further use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- infertile females prior to IVF: females diagnosed with idiopathic or male factor infertility. Follicular fluid samples will be obtained from all females following ovarian stimulation. Mature oocytes will be collected 34-36 h after human chorionic gonadotropin injection. Clinical follow up after embryo transfer, if the outcome will be a positive pregnancy test or clinical pregnancy with a fetal heartbeat at ≥ 8 weeks, the follicular fluid samples will be classified into the pregnancy group (I). In the absence of pregnancy, the samples will be classified as non-pregnancy group (ӀӀ)

SUMMARY:
1. Investigate the expression levels of circ-0033392, miR-375, miR-1305, JAK2, and PTEN in follicular fluids of females candidate for IVF.
2. Correlate the expression levels of measured biomarkers to the pregnancy rate and live birth rate.
3. Correlate the expression levels of the measured biomarkers with the embryological outcome which is the oocyte maturity rate, fertilization rate, embryo cleavage rate and blastocyst formation rate and implantation rate.

DETAILED DESCRIPTION:
Approximately 15-20% of reproductive-aged couples are suffering from infertility worldwide, and many couples turn to in vitro fertilization and embryo transfer (IVF-ET) technique. This technique is a multi-step process involving controlled ovarian hyperstimulation (COH), oocyte recovery, in vitro fertilization, embryo cultivation, embryo selection, and embryo transfer.

The success of the IVF process is conditioned by the receptivity of endometrium, the selection of a competent embryo for transfer, and the determination of the window of implantation (WOI). The biggest causes of the negative outcome of the IVF process are poor embryo quality and low endometrial receptivity.

The implantation capacity of a morphologically high-quality embryo reaches only 50%, and the success rate of IVF may therefore still not exceed 30%.

The increased interest in assisted reproduction through IVF leads to an urgent need to identify biomarkers that reliably highly predict the success of pregnancy.

The current paradox is that multiple embryo transfer that may leads to severe obstetric and perinatal complications seems to be the most valid measure to secure high success rate in the majority of clinic centers. Therefore, to avoid multiple transfer of embryos, it is urgent to explore biomarkers for IVF prognosis to select high-quality oocytes and embryos.

CircRNA, as a new class of non-coding RNA, exhibits high stability, abundance, and tissue specificity. It participates in the process of gene translation into protein and interacts with RNA binding protein through sponging miRNA or directly binding with RNA-binding proteins, and even translating into proteins.

Researchers have shown that circRNAs play important roles in cancer through the circRNA-miRNA-mRNA regulatory axis, thus affecting the occurrence and development of cancer. Many studies have shown that circRNAs can regulate the occurrence and development of different kinds of diseases.

CircRNA-mediated regulation in the ovary has drawn more and more attention recently , the biological functions of circRNAs in the ovary are still largely unknown. Liu et al. reported altered circular RNA expression in patients with recurrent implantation failure (RIF).

CircRNAs are commonly used as diagnostic and prognostic biomarkers. However, the exact role of circRNAs in implantation remains largely unknown.

Has-circ-0033392 is one of three key circRNAs were found to be mainly involved in the regulation of actin filament organization, focal adhesion, and cadherin binding.

Cadherins are a group of membrane proteins involved in cell adhesion, they assure adhesion between adjacent cells by the homotypic interactions of cells exposing similar sets of cadherins at their surfaces, cadherins contribute to tissue integrity, regulating cell migration, cell differentiation and the control size of a specific cell population, folliculogenesis strictly depends on the contact of the surrounding granulosa cells (GCs) and the oocyte.

Embryo implantation also involves the adhesion of trophoblast cells to the epithelial layer of the endometrium, dependent on cell-cell adhesion molecule interactions. However, so far, there is no research about has-circ-0033392 on diseases published.

MicroRNAs (miRNAs), a class of small non-coding RNAs with -22 nucleotides in length, regulate a wide array of biological processes, including embryonic development and response to pathogens. The mature miRNAs negatively modulate protein translation by binding to the 3ˋ-untranslated region (3ˋ-UTR) of target mRNAs.

MicroR-375 is expressed in GCs and oocytes and targets genes that regulate follicular growth proliferation, spread and apoptosis of cumulus cells (CCs).

Overexpression of miR-375 blocked the ability to proliferate, increased the apoptosis rate of cumulus cells in cows, and suppressed estradiol production and follicular development in porcine GCs.

MiR-375 was elucidated to repress cell proliferation and enhance the apoptosis in bovine CCs via regulation of bone morphogenetic protein type II receptor (BMPR2), highlighting its involvement in oocyte maturation. MiR-375 was preferentially detected in SBM samples of implanted blastocysts compared with blastocysts that failed to implant.

Previous studies found that miR-1305 promote cell proliferation, migration, and invasion in cervical cancer. The expression of miR-1305 was upregulated in epithelial ovarian carcinoma and that has miR-1305 regulates cell cycle and cell apoptosis. Overexpression of hsa-miR-1305 increases cell apoptosis, while its knockdown reduces the number of apoptotic cells.

Binding miR-1305 with Wnt2, and enhancing the Wnt/β-catenin pathway to promotes cell proliferation, migration, invasion. Components of the WNT signaling pathway have been demonstrated to impact reproductive functions including regulation of follicle maturation.

MiR-1305 was found to be upregulated in RIF. However, there is still no report linking miR-1305 to RIF.

The Janus kinases (JAK) are part of the tyrosine kinase group of enzymes of which four members have been identified: JAK1, JAK2, JAK3 and TYK2 (Tyrosine kinase 2). JAK2 links to the intracellular domain of many cytokine receptors for signal transduction. When cytokines bind to JAK2 receptors, the phosphorylation of JAK2 leads to the phosphorylation of other intracellular molecules, mainly through the JAK2-STAT3 pathway, which ultimately leads to gene transcription, It plays an important role in cytokine signal transduction and regulation of cell growth and gene expression.

In preimplantation embryos, STAT3 is constitutively active during fetal stage and shown to be important for embryonic development. Previous study showed that JAK2 regulated the microfilaments aggregation during the mouse oocyte maturation..

JAK2-mediated sodium/hydrogen exchange activation regulated acute cell volume changes in the late single-cell stage of mouse preimplantation embryos. Dysregulation of cell volume in early preimplantation embryos may lead to embryonic development arrest.

JAK/STAT pathway also among the most important signaling pathways of endometrial angiogenesis and the implantation of the embryo.

PTEN (encoding phosphatase and tensin homolog) is a tumor suppressor gene functions to control cell growth, differentiation, and survival by regulating every phase of the cell cycle, PTEN is crucial for mammal reproduction, in which it functions as a mediator of apoptosis in GCs.

Apoptosis is closely involved with most of reproductive processes, including folliculogenesis, follicle selection, and atresia. Apoptosis in GCs has been closely associated with follicular atresia, and was suggested to impact the ovarian reserve in women undergoing IVF treatment.

PTEN mRNA levels were significantly decreased in CCs surrounding mature oocytes compared with immature oocytes and were overexpressed of in poor responders. Failed IVF outcomes might be related to the high PTEN transcript levels in GCs.

Aim of the Research:

1. Investigate the expression levels of circ-0033392, miR-375, miR-1305, JAK2, and PTEN in follicular fluids of females candidate for IVF.
2. Correlate the expression levels of measured biomarkers to the pregnancy rate and live birth rate.
3. Correlate the expression levels of the measured biomarkers with the embryological outcome which is the oocyte maturity rate, fertilization rate, embryo cleavage rate and blastocyst formation rate and implantation rate.

ELIGIBILITY:
Inclusion Criteria:

1. Females age <40 years with male factor or idiopathic infertility.
2. Females undergo embryo transfer of blastocysts after intracytoplasmic sperm injection (ICSI) or conventional in vitro fertilization (IVF)

Exclusion Criteria:

1. Patients with structural and tissue abnormalities or infectious etiologies in the uterus and adnexa
2. Women with risk factors or diseases that could influence oocyte quality, such as women with body mass index ≥35 kg/m2, a diagnosis of polycystic ovarian syndrome or endometriosis or diminished ovarian reserve.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: females prior to IVF from attendants of IVF unit of Women's Health Hospital, Assiut university hospital, Assiut university.
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
levels of biomarkers | at time of egg retrieval
  Measure the expression of circ-0033392, miR-375, miR-1305, JAK2 and PTEN in follicular fluid samples from females prior to IVF.
Correlate biomarkers | ≥ 8 weeks after embryo transfer and follow up of pregnant females until delivery
  Correlate the expression levels of measured biomarkers to the pregnancy rate and live birth rate.

SECONDARY OUTCOMES:
Correlate biomarkers with embryological outcomes | at time of oocyte retrieval until embryo transfer
  Correlate the expression levels of the measured biomarkers with the embryological outcome which is the oocyte maturity rate, fertilization rate, embryo cleavage rate and blastocyst formation rate and implantation rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Biochemistry and Molecular Biology Department, Faculty of Medicine, Assuit University, Assuit, Egypt., Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Demographic and clinical data will include: Age (years), Body mass index, Number of previous pregnancies, previous live birth , previous abortion , Number of oocyte retrieved, Number of previous IVF attempts, Cause of infertility and Duration of infertility (years)
Supporting Information: Study Protocol